CLINICAL TRIAL: NCT01543685
Title: A Phase 3, Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Active- and Placebo-Controlled Study of Indomethacin [Test] Capsules for the Treatment of Acute Postoperative Pain After Bunionectomy
Brief Title: Study of Indomethacin Capsules to Treat Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND3-08-04b
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Other Acute Postoperative Pain
MeSH Terms: interventions — Indomethacin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Indomethacin 40 mg TID (Experimental)
  Interventions: Drug: Indomethacin
- Indomethacin 40 mg BID (Experimental)
  Interventions: Drug: Indomethacin
- Indomethacin 20 mg TID (Experimental)
  Interventions: Drug: Indomethacin
- Celecoxib 200 mg (Active Comparator)
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin — 40 mg TID capsules
  Arms: Indomethacin 40 mg TID
Drug: Indomethacin — 40 mg BID capsules
  Arms: Indomethacin 40 mg BID
Drug: Indomethacin — 20 mg TID capsules
  Arms: Indomethacin 20 mg TID
Drug: Celecoxib — 200 mg capsules
  Arms: Celecoxib 200 mg
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Indomethacin [Test] Capsules are safe and effective for the treatment of postoperative bunionectomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 65 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Has undergone primary, unilateral, first metatarsal bunionectomy with no additional collateral procedures
* Patient must be willing to stay at the study site ≥ 72 hours

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Clark, DPM, Principal Investigator — Premier Research Group Limited; Michael Golf, DPM, Principal Investigator — Premier Research Group Limited; Ira Gottlieb, DPM, Principal Investigator — Chesapeake Research Group, LLC; Kyle Patrick, DO, Principal Investigator — Premier Research Group Limited
Locations (4):
- United States (4):
  - Premier Research Group Limited, Phoenix, Arizona
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Premier Research Group Limited, Austin, Texas
  - Premier Research Group Limited, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Indomethacin 40 mg TID: Indomethacin : 40 mg TID capsules
- Indomethacin 40 mg BID: Indomethacin : 40 mg BID capsules
- Indomethacin 20 mg TID: Indomethacin : 20 mg TID capsules
- Celecoxib 200 mg: Celecoxib : 200 mg capsules
- Placebo: Placebo : Capsules
Period: Overall Study
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Started | 93 | 91 | 91 | 93 | 94
Completed | 90 | 88 | 89 | 93 | 90
Not Completed | 3 | 3 | 2 | 0 | 4
Not completed — Lack of Efficacy | 1 | 2 | 2 | 0 | 2
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib 200 mg | Indomethacin 20 mg TID | Indomethacin 40 mg BID | Indomethacin 40 mg TID | Placebo | Total
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94 | 462
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.3) | 41.5 (13.4) | 41.4 (12.4) | 41.5 (11.4) | 40.4 (13.3) | 41.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 79 | 72 | 79 | 77 | 384
  Male | 16 | 12 | 19 | 14 | 17 | 78
Region of Enrollment [Number; unit: participants]
  United States | 93 | 91 | 91 | 93 | 94 | 462

OUTCOME MEASURES:

1. Primary Outcome: The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale From 0 to 48 Hours After Trial Entry (VASSPID-48)
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  The VAS summed pain intensity difference (VASSPID) is calculated as the sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0 - 48 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
mm*hour | 508.2 (1125.6) | 329.8 (903.3) | 377.3 (1045.1) | 280.5 (799.8) | 69.4 (364.3)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = 441.8, 95% CI 2-sided [187.1 to 696.5], Standard Error of Mean 129.6
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.046, ANCOVA; Difference in Least Squares Mean = 260.2, 95% CI 2-sided [4.1 to 516.3], Standard Error of Mean 130.3
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA; Difference in Least Squares Mean = 312.7, 95% CI 2-sided [56.6 to 568.9], Standard Error of Mean 130.4
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.103, ANCOVA; Difference in Least Squares Mean = 211.6, 95% CI 2-sided [-43.1 to 466.2], Standard Error of Mean 129.6

2. Secondary Outcome: VASSPID-4. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 4 Hours After Trial Entry.
Description: as for outcome 1
Time Frame: 0 - 4 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
mm*hour | 30.7 (74.9) | 29.8 (70.8) | 17.9 (57.1) | 20.4 (54.6) | 8.9 (38.3)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.013, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.014, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.211, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.098, t-test, 2 sided

3. Secondary Outcome: VASSPID-8. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 8 Hours After Trial Entry.
Description: as for outcome 1
Time Frame: 0 - 8 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
mm*hour | 64.1 (144.6) | 55.4 (132.4) | 45.7 (122.7) | 37.2 (97.4) | 12.0 (49.9)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.028, t-test, 2 sided

4. Secondary Outcome: VASSPID-24. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 24 Hours After Trial Entry
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  The VAS summed pain intensity difference (VASSPID) is calculated as a time-weighted sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0 - 24 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
mm*hour | 226.9 (500.9) | 158.3 (405.2) | 176.9 (469.6) | 119.4 (329.6) | 28.3 (132.1)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.015, t-test, 2 sided

5. Secondary Outcome: Total Pain Relief (TOTPAR) Over 0 to 4 Hours (TOTPAR-4).
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 16 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 4 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
units on a scale*hour | 2.5 (3.6) | 2.1 (3.4) | 1.7 (2.9) | 1.8 (2.8) | 1.2 (2.1)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.022, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.146, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.071, t-test, 2 sided

6. Secondary Outcome: TOTPAR-8. Total Pain Relief (TOTPAR) Over 0 to 8 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 32 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 8 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
units on a scale*hour | 4.5 (7.4) | 3.4 (6.3) | 3.4 (6.3) | 3.0 (5.6) | 1.5 (2.9)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.010, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

7. Secondary Outcome: TOTPAR-24. Total Pain Relief (TOTPAR) Over 0 to 24 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 96 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 24 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
units on a scale*hour | 13.4 (26.4) | 8.9 (20.4) | 10.0 (23.0) | 7.7 (18.1) | 2.6 (8.8)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided

8. Secondary Outcome: TOTPAR-48. Total Pain Relief (TOTPAR) Over 0 to 48 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 192 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 48 hours
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Celecoxib 200 mg | Placebo
Number analyzed (Participants) | 93 | 91 | 91 | 93 | 94
units on a scale*hour | 29.3 (59.8) | 17.8 (45.6) | 19.6 (49.3) | 16.4 (43.2) | 5.2 (22.9)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.020, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.012, t-test, 2 sided
Statistical Analysis 4: Comparison: Celecoxib 200 mg vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Celecoxib 200 mg | Indomethacin 20 mg TID | Indomethacin 40 mg BID | Indomethacin 40 mg TID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/91 | 1/91 | 0/93 | 0/94
Other Adverse Events (participants affected / at risk) | 68/93 | 69/91 | 74/91 | 66/93 | 71/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 200 mg (N=93) | Indomethacin 20 mg TID (N=91) | Indomethacin 40 mg BID (N=91) | Indomethacin 40 mg TID (N=93) | Placebo (N=94)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 200 mg (N=93) | Indomethacin 20 mg TID (N=91) | Indomethacin 40 mg BID (N=91) | Indomethacin 40 mg TID (N=93) | Placebo (N=94)
Nausea (Gastrointestinal disorders) | 30 | 29 | 24 | 30 | 34
Dizziness (Nervous system disorders) | 7 | 6 | 14 | 12 | 16
Vomiting (Gastrointestinal disorders) | 3 | 10 | 7 | 5 | 13
Post procedural edema (Injury, poisoning and procedural complications) | 25 | 23 | 22 | 24 | 31
Headache (Nervous system disorders) | 5 | 11 | 13 | 12 | 7
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 8 | 6 | 13 | 5 | 6
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 1 | 3 | 0
Presyncope (Nervous system disorders) | 2 | 1 | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No